CLINICAL TRIAL: NCT04318613
Title: Antibiograms of Intensive Care Units at an Egyptian Tertiary Care Hospital
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Sherif M. S. Mowafy, Lecturer of anesthesia and surgical intensive care, Zagazig University
Other Study IDs: 5944-5-3-2020
Record Dates: First submitted 2020-03-18; First posted 2020-03-24 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The burden of antimicrobial resistance is high in ICUs and antibiotic therapy must continue to be used to improve health and save lives. However, the overuse or inappropriate use of antibiotics across the spectrum of healthcare and in the community is a leading cause of preventable antibiotic resistance development. Several achievements in medicine depend on effective antibiotic therapy and we need to preserve antibiotics to protect future generations. ICU physicians should have regularly updated antibiograms in order to guide appropriate decisions about the choice of empirical antibiotics when waiting for culture results. The appropriate selection of empirical antibiotic therapy should be guided by ICU-specific antibiogram.

DETAILED DESCRIPTION:
Hospital Acquired Infections (HAIs) surveillance at the local and national levels is an essential component of its control and prevention. The highest prevalence of HAIs is in Intensive care units (ICUs) and it is associated with considerable negative impact on the patients' outcome with a marked increase in the treatment costs. Therefore, early appropriate antibiotic therapy is a fundamental part of the treatment of these patients and it can be lifesaving. However, bacteria are becoming more resistant with alarming rates of antibiotic resistance worldwide.

Antibiotic resistance is part of a broader threat called antimicrobial resistance (AMR) that includes resistance to medicines used to treat all types of infections, including those caused by bacteria, parasites, and fungi. ICUs are considered the epicenter of AMR development due to the severity of critical illness, patients are at high risk of becoming infected through the use of invasive devices (e.g. endotracheal tubes, vascular and urinary catheters), and the extensive antibiotic use with variable infection control practices. Consequently, management of infections in ICU is a growing challenge and ICU physicians should have regularly updated antibiograms in order to guide appropriate decisions about the choice of empirical antibiotics when waiting for culture results Antibiograms are reports that summarize the information of bacterial antibiotic susceptibility rates within a single facility over the duration of one calendar year. They are used in tracking bacterial resistance and guiding empirical antibiotics prescription within the facility.

With the high burden of AMR and the ample variety between ICUs in the prevalence of micro-organisms and their antibiotic susceptibility, it is crucial that the selection of empirical antibiotic therapy should be guided by ICU-specific antibiogram. Also, the emerging trends in bacterial resistance at the local level should be monitored regularly.

The aim of this study is to find out the prevalence and types of pathogens and to determine their antibiotic susceptibility and resistance in different ICUs of an Egyptian tertiary care hospital (Zagazig University Hospitals).

ELIGIBILITY:
Inclusion Criteria:

* First isolate culture /patient .
* Only species with ≽ 30 isolates
* Diagnostic isolates
* Verified final results
* Routinely tested antimicrobial agents

Exclusion Criteria:

* Duplicate bacterial isolates
* Surveillance culture and screening isolates
* Reported Intermediate sensitivity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data was collected from all routine bacterial cultures in Zagazig University Hospitals' ICUs (emergency, surgical, medical, pulmonary, coronary, neonatal, and pediatric ICUs) over a one-year period from 1 /1/ 2019 to 31/12/ 2019.
Sampling Method: Probability Sample
Enrollment: 45221 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of micro-organisms at an Egyptian Tertiary Care Hospital | one year
  the prevalence and types of micro-organisms in Zagazig University Hospitals' ICUs by using data record base.
generation of ICU specific antibiogram | one year
  prepare and interprete antibiograms to guide empirical antibiotics prescription at ICUs of zagazig university hospitals by data record base cross sectional study
the incidence of antibiotic susceptibility and resistance pattern of these micro-organisms | one year
  the incidence of each antibiotic susceptibility and resistance pattern of micro-organisms at Zagazig University Hospitals' ICUs by record base study.

CONTACTS AND LOCATIONS:
Overall Officials: Sherif M Mowafy, MD, Principal Investigator — Anesthesia and Surgical Intensive Care Department, Faculty of Medicine, Zagazig University; Essamedin M Negm, MD, Study Director — Anesthesia and Surgical Intensive Care Department, Faculty of Medicine, Zagazig University; Ahmad A Mohammed, MD, Principal Investigator — Clinical Pathology Department, Faculty of Medicine, Zagazig University; Tarek H Hassan, MD, Principal Investigator — Chest Department, Faculty of Medicine, Zagazig University; Marwa G Amer, Master, Principal Investigator — Clinical Pathology Department, Faculty of Medicine, Zagazig University; Ahmed E Tawfik, Bachelor, Principal Investigator — Clinical pharmacist, Zagazig University Hospitals
Locations (1):
- Emergency, Surgical Intensive Care Units,medical, pulmonary, coronary, neonatal, and pediatric ICUs-Zagazig University Hospitals, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data that underlie results in the publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: the individual participant data and any additional supporting information will become available starting 6 months after publication.
Access Criteria: by contacting the study director

REFERENCES:
- [Background] Vincent JL, Rello J, Marshall J, Silva E, Anzueto A, Martin CD, Moreno R, Lipman J, Gomersall C, Sakr Y, Reinhart K; EPIC II Group of Investigators. International study of the prevalence and outcomes of infection in intensive care units. JAMA. 2009 Dec 2;302(21):2323-9. doi: 10.1001/jama.2009.1754. PMID 19952319
- [Background] van Hauwermeiren E, Iosifidis E, Karki T, Suetens C, Kinross P, Plachouras D. Development of case vignettes for assessment of the inter-rater variability of national validation teams for the point prevalence survey of healthcare-associated infections and antimicrobial use in European acute care hospitals. J Hosp Infect. 2019 Apr;101(4):455-460. doi: 10.1016/j.jhin.2019.01.018. Epub 2019 Jan 23. PMID 30682398
- [Background] Law T, Chibabhai V, Nana T. Analysis and comparison of cumulative antibiograms for the Charlotte Maxeke Johannesburg Academic Hospital adult intensive care and high-care units, 2013 and 2017. S Afr Med J. 2019 Dec 12;110(1):55-64. doi: 10.7196/SAMJ.2019.v110i1.13841. PMID 31865944
- [Background] Vincent JL, Bassetti M, Francois B, Karam G, Chastre J, Torres A, Roberts JA, Taccone FS, Rello J, Calandra T, De Backer D, Welte T, Antonelli M. Advances in antibiotic therapy in the critically ill. Crit Care. 2016 May 17;20(1):133. doi: 10.1186/s13054-016-1285-6. PMID 27184564
- [Background] Campion M, Scully G. Antibiotic Use in the Intensive Care Unit: Optimization and De-Escalation. J Intensive Care Med. 2018 Dec;33(12):647-655. doi: 10.1177/0885066618762747. Epub 2018 Mar 13. PMID 29534630
- [Background] Brusselaers N, Vogelaers D, Blot S. The rising problem of antimicrobial resistance in the intensive care unit. Ann Intensive Care. 2011 Nov 23;1:47. doi: 10.1186/2110-5820-1-47. PMID 22112929
- [Background] Hughes MA, Dosa DM, Caffrey AR, Appaneal HJ, Jump RLP, Lopes V, LaPlante KL. Antibiograms Cannot Be Used Interchangeably Between Acute Care Medical Centers and Affiliated Nursing Homes. J Am Med Dir Assoc. 2020 Jan;21(1):72-77. doi: 10.1016/j.jamda.2019.07.016. Epub 2019 Sep 16. PMID 31537479
- [Background] Kollef MH, Bassetti M, Francois B, Burnham J, Dimopoulos G, Garnacho-Montero J, Lipman J, Luyt CE, Nicolau DP, Postma MJ, Torres A, Welte T, Wunderink RG. The intensive care medicine research agenda on multidrug-resistant bacteria, antibiotics, and stewardship. Intensive Care Med. 2017 Sep;43(9):1187-1197. doi: 10.1007/s00134-017-4682-7. Epub 2017 Feb 4. PMID 28160023
- [Background] Cheesbrough M. District laboratory practice in tropical countries part II. 2. NewYork: Cambridge University Press; 2006.
- [Background] Clinical and Laboratory Standards Institute. Performance Standards for Antimicrobial Susceptibility Testing; 26th Edition. Wayne, PA: Clinical and Laboratory Standards Institute; 2016. CLSI document M100-S26.
- [Background] Magiorakos AP, Srinivasan A, Carey RB, Carmeli Y, Falagas ME, Giske CG, Harbarth S, Hindler JF, Kahlmeter G, Olsson-Liljequist B, Paterson DL, Rice LB, Stelling J, Struelens MJ, Vatopoulos A, Weber JT, Monnet DL. Multidrug-resistant, extensively drug-resistant and pandrug-resistant bacteria: an international expert proposal for interim standard definitions for acquired resistance. Clin Microbiol Infect. 2012 Mar;18(3):268-81. doi: 10.1111/j.1469-0691.2011.03570.x. Epub 2011 Jul 27. PMID 21793988